CLINICAL TRIAL: NCT07283614
Title: Impact of Preoperative Ocular Hypotony on Refractive Predictability After Phacovitrectomy for Rhegmatogenous Retinal Detachment
Brief Title: Ocular Hypotony and Refractive Predictability in RRD Surgery
Acronym: HYP-RRD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kazakh Eye Research Institute (Network)
Responsible Party: Principal Investigator, Kairat Ruslanuly, Dr, Kazakh Eye Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-194-2024
Record Dates: First submitted 2025-12-04; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Rhegmatogenous Retinal Detachment; Hypotony Ocular
Keywords: Rhegmatogenous Retinal Detachment; Hypotony Ocular; vitreoretinal sugery; cataract surgery; intraocular lens calculation; refractive assessment
MeSH Terms: conditions — Ocular Hypotension | interventions — Lens Implantation, Intraocular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RRD Patients with Ocular Hypotony (Active Comparator): Patients with primary rhegmatogenous retinal detachment (RRD) and preoperative ocular hypotony, defined as Goldmann intraocular pressure (IOP) ≤ 7 mmHg, undergoing combined phacoemulsification and IOL implantation, pars plana vitrectomy with silicone oil tamponade.
  Silicone oil is planned to be removed approximately 3 months after the initial combined surgery and detailed refractive assessment is performed 1 month after silicone oil removal. This cohort is used to evaluate the impact of preoperative hypotony on axial length measurements, refractive predictability (MAE, % within ±0.50 D), and visual outcomes.
  Interventions: Procedure: Combined Phacovitrectomy with Intraocular Lens Implantation and Silicone Oil Tamponade; Procedure: Silicone Oil Removal
- RRD patients with normal IOP (Active Comparator): Patients with primary rhegmatogenous retinal detachment (RRD) and normal preoperative IOP (> 7 mmHg) undergoing the same combined phacovitrectomy with IOL implantation and silicone oil tamponade.
  Silicone oil is planned to be removed approximately 3 months after the initial combined surgery and detailed refractive assessment is performed 1 month after silicone oil removal. This cohort serves as the comparison group for the hypotony arm to determine whether normal preoperative IOP is associated with more accurate axial length measurements, better refractive predictability, and comparable or superior visual outcomes.
  Interventions: Procedure: Combined Phacovitrectomy with Intraocular Lens Implantation and Silicone Oil Tamponade; Procedure: Silicone Oil Removal

INTERVENTIONS:
Procedure: Combined Phacovitrectomy with Intraocular Lens Implantation and Silicone Oil Tamponade — Standardized single-stage clear corneal phacoemulsification with IOL implantation is combined with three-port 25-gauge pars plana vitrectomy, fluid-air exchange, endolaser photocoagulation, and silicone oil tamponade for rhegmatogenous retinal detachment.
  After cataract extraction and IOL placement, pars plana vitrectomy is performed with fluid-air exchange to reattach the retina, endolaser photocoagulation around retinal breaks, and tamponade with silicone oil.
Procedure: Silicone Oil Removal — Silicone oil removal is performed approximately 3 months after the initial combined phacovitrectomy. Three-port 25-gauge pars plana access and pressure-controlled fluid-silicone exchange with balanced salt solution to completely remove silicone oil from the vitreous cavity. At the end of surgery, sclerotomies are sutured.

SUMMARY:
This study evaluates how preoperative ocular hypotony (Goldmann IOP ≤ 7 mmHg) affects refractive predictability, axial length measurements, and visual outcomes in patients undergoing combined phacovitrectomy with silicone oil for rhegmatogenous retinal detachment.

DETAILED DESCRIPTION:
This observational cohort study is designed to evaluate the impact of preoperative ocular hypotony (defined as Goldmann IOP ≤ 7 mmHg) on refractive outcomes, biometry parameters, and visual acuity after combined phacovitrectomy for RRD. All included eyes undergo standard 25-gauge pars plana vitrectomy with cataract extraction with IOL implantation, endolaser photocoagulation, and silicone oil tamponade.

The study population consists of eyes with primary RRD and stratified into two cohorts according to preoperative IOP:

Hypotony group - eyes with Goldmann IOP ≤ 7 mmHg; Control group - eyes with normal preoperative IOP .

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of primary rhegmatogenous retinal detachment (RRD);
2. Single-stage combined phacovitrectomy with clear corneal phacoemulsification with IOL implantation and 25G pars plana vitrectomy with silicone oil tamponade in the study eye;

4. Preoperative intraocular pressure (IOP) in the study eye measured by Goldmann applanation tonometry: Hypotony group: IOP ≤ 7 mmHg Normotony group: IOP > 7 mmHg 5. Planned silicone oil removal approximately 3 months after the initial combined surgery and ability to attend follow-up for refractive assessment 1 month after silicone oil removal; 6. Age (e.g., ≥18 years) and ability to provide informed consent;

Exclusion Criteria:

1. Previous intraocular surgery in the study eye;
2. Secondary or complex RRD associated with ocular trauma, uveitis or other active intraocular inflammation, proliferative diabetic retinopathy or other advanced vascular retinopathies, significant ocular malformations or congenital anomalies of the globe or posterior segment, pre-existing advanced glaucoma or uncontrolled ocular hypertension, or other optic nerve pathology that could confound visual and refractive outcomes, corneal opacity, significant corneal irregularity, or media opacity precluding reliable biometry or accurate axial length measurement in the study eye, systemic diseases or autoimmune conditions with known ocular involvement that may affect the retina, choroid, or refraction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-12-08 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-10-17 (Estimated)

PRIMARY OUTCOMES:
Mean Absolute Error (MAE) of Postoperative Refraction | 1 month after silicone oil removal
  Mean Absolute Error between the target refraction predicted by preoperative IOL power calculation and the achieved postoperative spherical equivalent refraction, calculated in diopters for each eye. Percentage of eyes in each group with an Mean Absolute Error ≤ ±0.50 diopters between the target refraction and the achieved postoperative spherical equivalent refraction.

SECONDARY OUTCOMES:
Axial Length Measurement | 1 month after silicone oil removal
  Difference between preoperative and postoperative axial length measurements, and its association with preoperative IOP status.
Best-Corrected Visual Acuity | 3 months after combined surgery, 1 month after silicone oil removal
  Best-Corrected Visual Acuity measured in Logarithm of the Minimum Angle of Resolution (LogMAR) units using standard visual acuity charts and compared between hypotony and normotony groups after surgery and silicone oil removal

CONTACTS AND LOCATIONS:
Locations (1):
- Kazakh Eye Research Institute, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: Undecided